CLINICAL TRIAL: NCT00181974
Title: Efficacy of a Fibrin Sealant in Burn Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Robert L. Sheridan, Surgeon, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Not sponsored
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Burns
Keywords: burns; hemostasis; skin graft; Surgical Hemostasis; Grafting, Skin
MeSH Terms: conditions — Burns

INTERVENTIONS:
Drug: Tisseel Fibrin Sealant

SUMMARY:
The purpose of this study is to determine the effectiveness of a fibrin glue in burn surgery with respect to hemostasis and skin graft fixation.

DETAILED DESCRIPTION:
Burn patients require extensive split-thickness skin grafting operations. These operations necessitate excision of burn wounds and the procurement of autografts. Both of these result in bleeding open wounds. Fibrin sealants may be of benefit in three aspects of burn surgery:

1. as a hemostatic agent on excised burns,
2. as a hemostatic agent on donor sites, and
3. as a method of fixation of skin grafts to wounds.

Skin grafts are routinely secured with surgical staples. Patients with large burns will commonly have hundreds, even thousands of staples used during the course of their care. Problems associated with the use of surgical staples include:

1. discomfort upon removal and
2. staples become deeply embedded in the tissue.

If effective in securing skin grafts, fibrin glue would directly benefit burn patients by decreasing the number of staples required, and thereby decreasing the number of retained staples. Fibrin sealant is produced from human fibrinogen and human thrombin from pooled plasma that is virally inactivated by a two-stage heating process.

Subjects will serve as their own control. They will have an area of their wound treated with the fibrin sealant and another area treated with the standard of care. Both areas will be compared for hemostasis, skin graft fixation, wound healing, and cosmetic outcome.

ELIGIBILITY:
Inclusion Criteria:

* Requires skin grafting of an acute or reconstructive burn wound.

Exclusion Criteria:

* Active disseminated intravascular coagulation (DIC) or known hypersensitivity to bovine protein.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2000-03; Primary Completion 2007-02 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
initial wound hemostasis
initial donor site hemostasis
initial graft fixation
percent graft take at 1 week
outcome and cosmetic appearance at routine intervals up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Sheridan, M.D., Principal Investigator — Shriners Burns Hospital
Locations (1):
- Shriners Burns Hospital, Boston, Massachusetts, United States